CLINICAL TRIAL: NCT06361537
Title: Prospective, Multicenter, Randomized, Double-blind, Parallel Group, Placebo- Controlled, Efficacy and Safety Phase 3 Study of an Intravenous Human Plasma- Derived C1 Esterase Inhibitor (C1-INH) Concentrate in Participants With Congenital C1-INH Deficiency for the Treatment and Pre-procedure Prevention of Acute Hereditary Angioedema Attacks
Brief Title: Study of IV Human Plasma-derived C1 Esterase Inhibitor Concentrate in Patients With Congenital C1-INH Deficiency for Treatment and Pre-procedure Preventing of Acute Hereditary Angioedema Attacks
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CONE-02
Record Dates: First submitted 2024-01-11; First posted 2024-04-12 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Acute Hereditary Angio Edema
Keywords: Edema; Swelling; Angio Edema; Hereditary; Congenital Angioedema
MeSH Terms: conditions — Edema; Angioedema

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- OCTA-C1-INH (Experimental): OCTA-C1-INH injection, 20IU/kg BW after first qualifying attack. Treatment to be administered to blinded as well as open-label subjects.
  Interventions: Drug: OCTA-C1-INH
- Placebo (Placebo Comparator): 0.1 mL/kg BW 0.9% sodium chloride solution injection after first qualifying attack. Only blinded subjects to receive.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: OCTA-C1-INH — OCTA-C1-INH is a stable, sterile, virus-inactivated, nano-filtered, highly purified concentrate of human C1-INH prepared from pooled human plasma. After reconstitution in 2.5mL water for injection, the solution can be administered as a slow IV injection. OCTA-C1-INH is given as a dose of 20 IU/kg body weight (BW)
  Arms: OCTA-C1-INH
Other: Placebo — 0.1 mL/kg BW 0.9% sodium chloride injection
  Arms: Placebo

SUMMARY:
Prospective, multicenter, randomized, double-blind, parallel group, placebo- controlled, efficacy and safety phase 3 study of an intravenous human plasma- derived C1 esterase inhibitor (C1-INH) concentrate in participants with congenital C1-INH deficiency for the treatment and pre-procedure prevention of acute hereditary angioedema attacks

ELIGIBILITY:
Inclusion Criteria:

1. Is at least 18 years of age (applicable for 1st study phase) or is at least 2 years of age (applicable for 2nd study phase)
2. Has confirmed diagnosis of HAE type I or II
3. Has had at least 3 moderate or severe HAE attacks (excluding extremity attacks) in the last 3 months before the Screening Visit. For participants ≥2 and ≤12 years of age, has had at least 1 moderate or severe HAE attack (excluding extremity attacks) in the last 6 months before Screening Visit
4. Has a documented congenital C1-INH functional activity <50% with or without C1-INH deficiency and C4 antigen level below the laboratory reference range
5. Participant or the participant's legally authorized representative(s) has signed informed consent (as required by local law), with the assent of participants legally capable of providing it, as applicable
6. States willingness to comply with all study procedures and availability for the duration of the study
7. If the participant is of childbearing potential (CBP), has a negative pregnancy test and must have been using a highly effective method of contraception and continue to do so until at least 2 weeks after their last dose (for both blinded and open-label doses of IMP). Not of CBP is defined as surgically sterilized (hysterectomy, bilateral oophorectomy) or who are postmenopausal (defined as women with no menses for 12 months without an alternative medical cause). Highly effective methods of contraception:

   * Combined hormonal contraception (estrogens and progesterone) methods such as oral, implantable, intravaginal, injectable, or transdermal contraceptives at a stable dose for a minimum of 1 full cycle (hormonal contraceptives must inhibit ovulation) and for at least 4 weeks before screening
   * Progesterone only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
   * Intrauterine device
   * Intrauterine hormone-releasing system inserted at least 4 weeks before screening
   * Bilateral tubal ligation/occlusion or vasectomized partner (with surgical success confirmed by medical assessment) OR Agrees to abstain from heterosexual intercourse during study participation and to use a highly effective contraceptive (as described above) as backup if they become sexually active during the study. Abstinence is only acceptable if this is the participant's usual lifestyle. Periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method are not acceptable methods of contraception
   * Note: If a participant of CBP has a positive or suspected positive urine pregnancy test within 72 hours prior to treatment, a serum pregnancy test will be required
   * Male participants must not plan to father a child or donate sperm for 90 days after their last dose of study drug (for both blinded and open-label doses of the IMP). However, there are no official contraception requirements for male participants during the study.

Inclusion Criteria for IMP Dosing for QAT:

1. Has confirmed QAT per definition criteria
2. Has a swelling episode that is new and not the continuation of a previous HAE attack

Exclusion Criteria:

1. Has a history of clinically relevant antibody development against C1-INH
2. Has a medical history consistent with Type 3 HAE (i.e., onset at age above 40 year, no family history, no known HAE mutation, low C1q level in plasma)
3. Has a history of allergic reaction to C1-INH or other blood/plasma product
4. Has a history of B-cell malignancy that was unresolved in the past 5 years
5. Has a narcotic and/or alcoholic addiction
6. Has participated in any other investigational drug evaluation within 30 days before screening
7. Is pregnant or breastfeeding
8. Has any clinically significant medical or psychiatric condition that, in the investigator's opinion would interfere with the participant's ability to participate in the study
9. Has a history of thromboembolic events (TEEs), myocardial infarction, unstable angina pectoris, critical aortic stenosis, cerebrovascular accident, transient ischemic attack, severe peripheral vascular disease, or disseminated intravascular coagulation within one year before screening
10. (applicable until IDMC review of the interim preliminary safety and efficacy data): has clinically significant derangement in measurements of cardiovascular status (i.e. uncontrolled arterial hypertension, cardiac insufficiency New York Heart Association (NYHA) class III-IV), pulmonary status (i.e., COPD GOLD classification 3 and 4, severe asthma) and renal status (i.e., eGFR below 90 ml/min per 1.73 m2)

Exclusion Criteria for IMP Dosing for QAT:

1. Has received blood or a blood product for prophylactic or acute treatment with any C1-INH (Berinert®, Cinryze®, HAEgarda®, Ruconest®, etc.), non-biological bradykinin and kallikrein pathway inhibitors (e.g., ecallantide, icatibant, berotralstat), or treatment with tranexamic acid within 14 days before dosing with the IMP (or is not willing to abstain from these medications throughout the study)
2. started or changed hormone replacement therapy or selective estrogen receptor modulators (e.g., tamoxifen) within 14 days before IMP dosing
3. Started or changed androgen therapy (e.g. testosterone, dehydro- epiandrosterone/androstenedione, oxandrolone, danazol, stanozolol) within 14 days before IMP dosing or is not willing to maintain a stable dose throughout the study
4. Started or changed the dose of monoclonal antibodies e.g. lanadelumab within 11 weeks before dosing or not willing to maintain a stable dose throughout the study
5. Has used narcotic pain medications or non-opioid analgesics within 7 days before IMP dosing for a QAT
6. Has received OCTA-C1-INH within 14 days before IMP dosing

Exclusion Criteria for IMP Dosing for PK:

1. Has received blood or a blood product for prophylactic or acute treatment with any C1-INH (Berinert®, Cinryze®, HAEgarda®, Ruconest®, etc.), non-biological bradykinin and kallikrein pathway inhibitors (e.g., ecallantide, icatibant, berotralstat), or treatment with tranexamic acid within 14 days before dosing with the IMP (or is not willing to abstain from these medications throughout the study)
2. Is receiving hormone replacement therapy or selective estrogen receptor modulators (e.g., tamoxifen) and has had their dose changed within 14 days before IMP dosing
3. Is receiving or has received androgen therapy (e.g., testosterone, dehydroepiandrosterone/androstenedione, oxandrolone, danazol, stanozolol) IN ANY DOSE within 14 days before dosing
4. Started or changed the dose of monoclonal antibodies e.g lanadelumab within 11 weeks before dosing or not willing to maintain a stable dose throughout the study
5. Has used narcotic pain medications or non-opioid analgesics within 7 days before IMP dosing
6. Has received IMP within 14 days before IMP dosing
7. Has planned dental, medical, or surgical procedures during the PK Period that will require pre-procedural prevention

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Time (h) to beginning of unequivocal symptom relief at the defining site in blinded participants. | Within 4 hours after injection
  Patient will rate symptom relief for the defining attack site (site of swelling or pain) from 15 minutes after start of the IMP injection every 15 minutes over 4 hours. Unequivocal relief is defined as having 3 consecutive reports of "absent now but present before," "absent now and absent before", or "present, symptoms better" on the 5-grade SRRS.
  This measure will also be used for the secondary outcomes in a different context.

SECONDARY OUTCOMES:
Percentage of participants responding to treatment | within 4 hours after injection
  Percentage of patients responding to treatment, defined as beginning of unequivocal symptom relief at the defining site within 4 hours after injection (once per participant after first qualifying attack in the study). Unequivocal relief is defined as having 3 consecutive reports of "absent now but present before," "absent now and absent before", or "present, symptoms better" on the 5-grade symptom relief rating.
Time to beginning of unequivocal symptom relief at all sites involved | Within 4 hours after injection
  Time to the beginning of unequivocal symptom relief at all sites involved within 4 hours after injection. Unequivocal relief is defined as having 3 consecutive reports of "absent now but present before," "absent now and absent before", or "present, symptoms better" on the 5-grade symptom relief rating.
Changes in symptom severity at the defining site by VAS severity rating | Within 4 hours after injection
  Changes in symptom severity at the defining site by visual analog scale (VAS) rating from pre-injection over 4 hours after injection. The VAS is a self-reported 0-100 pain and swelling rating scale.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (3):
  - Octapharma Research Site, Centennial, Colorado
  - Octapharma Research Site, Farmington Hills, Michigan
  - Octapharma Research Site, Toledo, Ohio
- Octapharma Research Site, Tirana, Albania
- Octapharma Research Site, Rosario, Argentina
- Octapharma Research Site, Yerevan, Armenia
- Octapharma Research Site, Sofia, Bulgaria
- Mexico (2):
  - Octapharma Research Site, Lima
  - Octapharma Research Site, Mexico City
- Octapharma Research Site, Podgorica, Montenegro
- Octapharma Research Site, Lima, Peru
- Octapharma Research Site, Cluj-Napoca, Romania
- Octapharma Research Site, Kragujevac, Serbia
- Turkey (Türkiye) (4):
  - Octapharma Research Site, Ankara
  - Octapharma Research Site, Istanbul
  - Octapharma Research Site, Izmir
  - Octapharma Research Site, Sakarya
- Ukraine (2):
  - Octapharma Research Site, Kyiv
  - Octapharma Research Site, Lviv

IPD SHARING:
Plan to Share IPD: No